CLINICAL TRIAL: NCT01929499
Title: Efficacy of Adjuvant Immunotherapy With Cytokine-induced Killer Cells in Patients With Stage II/III Colon Cancer
Brief Title: Efficacy of Adjuvant Cytokine-induced Killer Cells in Colon Cancer
Acronym: CIKCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yanjuan Zhu (Other)
Responsible Party: Sponsor-Investigator, Yanjuan Zhu, Department of Oncology, Guangdong Provincial Hospital of Traditional Chinese Medicine
Organization: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIKCC
Record Dates: First submitted 2013-08-20; First posted 2013-08-28 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Colonic Neoplasms
Keywords: Colon cancer; Cytokine-induced killer cells; Adjuvant immunotherapy; Adjuvant chemotherapy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- synchronous CIK group (Experimental): After colectomy, patients will accept chemotherapy combined with cytokine-induced killer cells (CIK) therapy synchronously for 6 months.
  For CapeOx regimen:
  3×109 CIK cells on days 1-3; Oxaliplatin 130mg/m2 on day 7; Capecitabine 1000mg/m2 twice daily on days 7-20; Repeat every 3 weeks for 6-8 cycles.
  For mFolfox6 regimen:
  Oxaliplatin 85mg/m2 IV over 2 hours on day 1; Leucovorin 400mg/m2 IV over 2 hours on day 1; 5-FU 400mg/m2 IV bolus on day 1, then 2400mg/m2 IV continuous infusion over 46-48 hous; 3×109 CIK cells on days 9-11; Oxaliplatin 85mg/m2 IV over 2 hours on day 15; Leucovorin 400mg/m2 IV over 2 hours on day 15; 5-fluorouracil (5-FU) 400mg/m2 IV bolus on day 15, then 2400mg/m2 IV continuous infusion over 46-48 hours; Repeat every 4 weeks for 5-6 cycles.
  Interventions: Biological: cytokine-induced killer cells
- sequence CIK group (Experimental): After colectomy, patients will accept adjuvant chemotherapy for 6 months, that is 6-8 cycles of CapeOX regimens (the same as those in arm A), or 10-12 cycles of mFolfox6 regimens(the same as those in arm A), followed by 6-8 cycles of cytokine-induced killer cells (CIK) therapy at least 2 weeks later.
  Interventions: Biological: cytokine-induced killer cells
- control group (No Intervention): After colectomy, patients will accept adjuvant chemotherapy for 6 months, that is 6-8 cycles of CapeOX regimens (the same as those in arm A), or 10-12 cycles of mFolfox6 regimens （the same as those in arm A）.

INTERVENTIONS:
Biological: cytokine-induced killer cells
  Other Names: CIK; cytokine induced killer cells
  Arms: sequence CIK group; synchronous CIK group

SUMMARY:
It has been reported that the immune status of patients with cancer were suppressed, especially those after surgery and adjuvant chemotherapy. Thus, immunotherapy may decrease the recurrence rate after surgery. CIK cells transfusion has been reported as an effect therapy in advanced cancers. In another retrospective study, investigators found that adjuvant CIK therapy would prolong the disease-free survival (DFS) for colorectal cancer patients.

The purpose of this study is to determine wether adjuvant immunotherapy with CIK cells in patients with colon cancer after operation will prolong DFS, and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Colon cancer in stage III or stage II with high risk after R0 resection
* Eastern Cooperative Oncology Group (ECOG) performance status was 0 - 1;
* Life expectancy of at least 3 months;
* Normal bone marrow, liver, renal, heart and lung function;
* Age between 18-80;
* Patients who provided written informed consent for this study

Exclusion Criteria:

* With uncontrolled other malignant tumors;
* With uncontrolled infection or tubercle bacillus (TB) or underlying diseases that were severe or life threatening;
* Patients who need to treat with radiotherapy;
* Patients who accepted other immunotherapy
* With sever mental disease or disease with central nervous system (CNS);
* With the history of organ transplantation, including bone marrow transplantation or stem cell transplantation;
* Patients with auto immune diseases;
* pregnant or lactating.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
DFS (Disease free survival) | Time elapsedelapsed from the date of surgery to either the date of recurrence or the date of last follow-up information,whichever come first, assessed up to 5 years.
  Patients who were recurrence free at the end of study or lost to follow-up were censored

SECONDARY OUTCOMES:
OS (overall survival) | Time elapsed from the date of surgery to either the date of death or the date of last follow-up information, whichever came first, assessed up to 5 years.
  Patients who were survival at the end of study or lost to follow-up were censored
Side effect | Up to 2 years
  Any undesirable secondary effect which occurs in addition to the desired therapeutic effect of CIK or chemotherapy, during the period from the first cycle of chemotherapy or CIK infusion to the end of study. The side effects were described according to the NCI-CTCAE (National Cancer Institute-Common Terminology Criteria for Adverse Events)
T lymphocyte subset | Up to 6 months
  During the period of CIK infusion
QoL (quality of life) | Up to 1 year
  During the period of chemotherapy and CIK infusion

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Zhang, MD, Principal Investigator — Guangdong Provincial Hospital of Chinese Medicine, China
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China